CLINICAL TRIAL: NCT05761210
Title: Characterization of Serum Proteome in Young Obese Subjects With Different Degrees of Liver Steatosis
Brief Title: Characterization of Serum Proteome in Young Obese Subjects (POSING)
Acronym: POSING
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C217
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Obesity; Proteome; Steatosis; Biomarkers
MeSH Terms: conditions — Obesity; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum/plasma samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases; subjects with steatosis
  Interventions: Diagnostic Test: Blood sample collection
- controls; subjects without steatosis
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Blood sample collection

SUMMARY:
With the project proposal we aim to identify serum markers for the characterization of steatosis in subjects affected by essential obesity at a young age. In this case the markers could be useful not only for the development of new diagnostic scores, or for combining them with diagnostic imaging technologies, but also for understanding the metabolic alterations according to the patient's gender, extremely important data in this disease to which only recently has biomedical research started.

DETAILED DESCRIPTION:
Experimental design The study includes a discovery phase in which a serum proteomic analysis of the subjects included in the study will be performed. This phase will make it possible to identify a small number of possible candidate markers, which will be validated in a subsequent phase with a greater number of subjects.

Patients:

In the discovery phase, 60 pubescent subjects (30 males and 30 females) will be taken into consideration. The subjects will be divided into two groups:

* control group including subjects with absence of steatosis, verified by ultrasound method according to standardized criteria [10,11], and with APRI score < 0.3;
* study group with subjects with the proven presence of steatosis using ultrasound techniques, and with APRI score > 0.50.

For each patient, the following variables will be considered in baseline conditions, i.e. at the time of sample collection.

* anthropometric parameters (height, weight, BMI, waist circumference);
* body composition (lean mass, fat mass), using the impedance measurement technique (BIA);
* levels of steatosis measured with ultrasound according to standard criteria
* blood chemistry parameters
* basic metabolism, using indirect calorimetry;
* biochemical parameters determining the metabolic syndrome (HDL cholesterol, triglycerides, blood sugar);
* biochemical parameters for the prediction of hepatic steatosis using surrogate markers (AST, ALT, GGT, platelets, alkaline phosphatase, albumin);
* blood pressure;
* concomitant hormonal therapies (growth hormone therapy, sex steroids, and/or l-thyroxine).

Serum collection Fasting blood samples will be collected by standard venipuncture into BD Vacutainer® serum separation tubes (BD - Plymouth PL6 7BP, UK) and centrifuged at 1900g at 4°C for 10 min and at 16,000g at 4°C for a further 10 min. The supernatants will be transferred to new tubes and subsequently frozen at -80°C for long-term storage.

Proteomic analysis Before the proteomic analysis, the presence of hemoglobin will be evaluated by spectrophotometer Beckman Coulter® DU®730 (Beckman Coulter, Brea, CA, USA) using the direct spectrophotometric method of Harboe with Allen correction: Hb ( g / L) = (167, 2 × A415 - 83.6 × A380 - 83.6 × A450) x 1/1000 × 1 / dilution in dH2O. The cut-off considered for serum will be 0.020 g/L.

For the proteomic characterization of serum, a new high-throughput omics technology based on the SomaLogic SOMAscan platform will be used. The system is based on the detection of SOMAmers (Slow Off-rate Modified Aptamers), which are aptameric forms of DNA with high affinity and specificity for the protein target. Furthermore, these aptamers are resistant to nucleotidase activity and demonstrate higher affinity than normal antibodies. The panel used in this study will allow us to evaluate 1500 protein targets that are involved in the development of metabolic diseases, are part of the general inflammatory response, and are of interest in the study of cardiovascular diseases and also in oncology.

In general, the sensitivity and performance of the test are comparable to that of a normal ELISA kit, with limits for quantification around 100 fM and detection of 40 fM, and the need for only 65 µL of the sample.

Validation The validation of 2 markers selected based on the significance and differential expression between the groups will be validated by the ELISA method. In this phase, each marker will be validated by determining its concentration in the serum of 60 subjects (included in the discovery phase) and in other 32 complementary subjects to reach the sample size useful for obtaining an appropriate statistical significance.

Furthermore, the experiments will be set up to include positive and negative controls and controls to check for inter-plate variability, as required by ELISA assay set-up procedures. Standard curves will be calculated to determine the absolute quantification of the markers of interest in serum.

ELIGIBILITY:
Inclusion Criteria:

* obesity (BMI SDS > 2)
* age range: 13-18

Exclusion Criteria:

- age < 13 years and > 18 years

Ages: 13 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Obese adolescents (BMI SDS > 2) with or without steatosis
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Identification of serum markers (proteomic analysis) for the characterization of steatosis in young subjects with essential obesity | Baseline
  Identification of serum markers (proteomic analysis)for the characterization of steatosis in young subjects with essential obesity

SECONDARY OUTCOMES:
Relationships between proteoma and body composition (evaluated throughout bioimpedentiometry) | Baseline
  Relationships between proteoma and body composition parameters (evaluated throughout bioimpedentiometry)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy